CLINICAL TRIAL: NCT04747795
Title: Early Administration of Vitamin C in Patients With Sepsis or Septic Shock in Emergency Departments: a Multicentre, Double Blinded, Randomized Controlled Trial: the C-EASIE Trial
Brief Title: Early Administration of Vitamin C in Patients With Sepsis or Septic Shock in Emergency Departments
Acronym: c-easie
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Federaal Kenniscentrum voor Gezondheidszorg, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S63213; 2020-001862-12 (EudraCT Number); KCE 19-1237 (Other Grant/Funding Number: Federaal kenniscentrum voor de gezondheidszorg (KCE))
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-09

CONDITIONS: Sepsis; Septic Shock; Sepsis, Severe
Keywords: Vitamin C; ascorbic acid; sepsis; septic shock; RCT
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care + placebo (Placebo Comparator): The 'standard care' group will receive intermittent infusion of normal saline (3 ampoules of 5 ml 9mg/ml normal saline diluted in 50 ml of normal saline, every 6 hours) during 4 days or until hospital discharge and is started within 6 hours after presentation (time of triage) in the ED.
  Interventions: Drug: Normal saline
- standard care + Vitamin C (Active Comparator): The 'standard care + Vitamin C' group will receive intermittent infusion of Vitamin C (3 ampoules of 500 mg/5ml Vitamin C diluted in 50 ml of normal saline, every 6 hours) during 4 days or until hospital discharge and is started within 6 hours after presentation (time of triage) in the ED.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — IV
  Other Names: Ascorbic Acid
  Arms: standard care + Vitamin C
Drug: Normal saline — IV
  Other Names: physiological serum; placebo
  Arms: standard care + placebo

SUMMARY:
In this clinical trial the effect of early administration of Vitamin C is investigated in patients admitted at the emergency department with sepsis or septic shock.

When a patient has sepsis, his/her body is causing damage to its own tissues and organs as result of an infection. This can lead to septic shock. The patient has a low blood pressure, his/her organs stop working and the patient may even die.

The aim of this trial is to investigate the efficiency of Vitamin C in sepsis and septic shock. Vitamin C is a vitamin present in various foods and has been approved as dietary supplement by the Belgian authorities. Over the years it has been proven that Vitamin C is very safe. In addition, several studies have shown that Vitamin C can also have a protective effect. It can reduce organ damage and increase survival rates. Although several studies suggest that Vitamin C can help fight sepsis, it is not yet used in practice. This Belgian trial, in which several hospitals participate, hopes to provide a clear answer to the question: "Should Vitamin C be administered to patients admitted in an emergency department with sepsis or septic shock?"

ELIGIBILITY:
Inclusion Criteria:

* Patient has a 'suspected infection': this requires the combination of antibiotic administration and body fluid cultures within the first 6 hours after Emergency Department presentation.
* Patient has a NEWS score ≥ 5.

Exclusion Criteria:

* Patient (≥18 years old) or legally authorized representative didn't provide informed consent. Delayed informed consent can be applied in cases where the patient is critically ill and no LAR is available.
* antibiotic administration as a single dose or as a prophylactic treatment.
* antibiotics administered without an accompanying body fluid culture according to the timeframe (within 6 hours after emergency department presentation).
* 'Do no intubate' or 'comfort measures only' status.
* Failure to randomize within 6 hours after Emergency Department presentation.
* Weight < 45 kg.
* Pregnant or breastfeeding.
* Known allergy for Vitamin C.
* Known history of oxalate nephropathy or hyperoxaluria.
* Known history of glucose-6-phosphate dehydrogenase deficiency.
* Known history of chronic iron overload due to iron storage and other diseases.
* The patient is already on IV steroids for a reason other than septic shock.
* Proven active COVID-19 infection (positive swab and/or CT scan positive for COVID-19 within 14 days prior to or at ED presentation).
* Participation in an interventional trial with an investigational medicinal product (IMP) or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score | 5 days
  Average post-baseline patient SOFA score, SOFA score range: 0-24, with 24 being the worst outcome (death)

SECONDARY OUTCOMES:
28-day mortality | 28 days
Maximum SOFA score | 5 days
  Maximum SOFA score measured during 5 intervention period. SOFA score ranging from 0 to 24, with 24 begin the worst outcome (death)
Length of hospital stay | 3 months
  Total length of hospital stay of the patient (including beyond intervention period)
Length of ICU stay | 3 months
  Total length of ICU stay of the patient (including beyond intervention period)
Duration Vasopressors | 5 days
  Total duration where vasopression is required (hours)
Dosage Vasopressors | 5 days
  Total dosage of Vasopressors required (mcg/kg/min)
need for Renal Replacement Therapy (RRT) | 5 days
  was RRT needed
duration of Renal Replacement Therapy (RRT) | 5 days
  total duration of RRT (hours)
Ventilator days | 3 months
  Total number of days the patient requires ventilator support (including beyond intervention period)
Steroids | 5 days
  Total dose of steroids given
Quality of life questionnaire (EQ-5D-5L) | 3 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Time to return to work | 3 months
  Time to return to work of the patient after ED admission (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Didier Desruelles, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (8):
- Belgium (8):
  - GasthuisZusters Antwerpen, Antwerp
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Centre Hospitalier Universitaire Saint-Pierre Bruxelles, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Université Libre de Bruxelles Erasme, Brussels
  - Universitaire Ziekenhuizen Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Algemeen Ziekenhuis Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vandervelden S, Cortens B, Fieuws S, Eegdeman W, Malinverni S, Vanhove P, Monsieurs K, Breuls J, Hubloue I, Stifkens F, Creteur J, Wauters L, Desruelles D; C-EASIE investigators. Early administration of vitamin C in patients with sepsis or septic shock in emergency departments: a multicenter, double-blind, randomized controlled trial: the C-EASIE trial. Crit Care. 2025 Apr 23;29(1):160. doi: 10.1186/s13054-025-05383-x. PMID 40269974
- [Derived] Vandervelden S, Wauters L, Breuls J, Fieuws S, Vanhove P, Hubloue I, Bartiaux M, Creteur J, Stifkens F, Monsieurs K, Desruelles D. Early administration of Vitamin C in patients with sepsis or septic shock in emergency departments: A multicenter, double blinded, randomized controlled trial: The C-EASIE trial protocol. PLoS One. 2021 Nov 5;16(11):e0259699. doi: 10.1371/journal.pone.0259699. eCollection 2021. PMID 34739527

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT04747795/SAP_000.pdf